CLINICAL TRIAL: NCT02802865
Title: Combined Letrozole and Clomid in Polycystic Ovary Syndrome: a Randomized Control Trial of Combination of Letrozole and Clomiphene Citrate or Letrozole Alone for the Treatment of Infertility in Women With Polycystic Ovary Syndrome
Brief Title: Combined Letrozole and Clomid in Women With Infertility and PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rachel Mejia (Other)
Responsible Party: Sponsor-Investigator, Rachel Mejia, Associate Fellow, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201606806
Record Dates: First submitted 2016-06-09; First posted 2016-06-16 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Polycystic Ovary Syndrome; Infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Clomiphene; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Letrozole (Active Comparator): Letrozole 2.5 mg orally for 5 days on cycle days 3-7
  Interventions: Drug: Letrozole
- Letrozole + Clomiphene (Experimental): Letrozole 2.5 mg orally for 5 days on cycle days 3-7 AND Clomid 50 mg orally for 5 days on cycle days 3-7
  Interventions: Drug: Clomiphene; Drug: Letrozole

INTERVENTIONS:
Drug: Clomiphene
  Other Names: clomid; clomiphene citrate
  Arms: Letrozole + Clomiphene
Drug: Letrozole
  Other Names: femara

SUMMARY:
This study evaluates the addition of clomid to letrozole for the treatment of infertility in women with polycystic ovary syndrome. Half of the participants will receive letrozole and clomid in combination, while the other half will receive letrozole alone.

DETAILED DESCRIPTION:
Letrozole and Clomid are both used for ovulation induction, but they have different mechanisms of action. Letrozole has been shown to be superior to clomid in achieving live birth rates in women with infertility and polycystic ovary syndrome. However, the combination of these medications has not been studied. This is a pilot study to evaluate if the combination treatment has improved efficacy as measured by ovulation rate.

This is a randomized controlled trial of letrozole versus letrozole and clomiphene citrate (CC) for one menstrual cycle. Women will be randomized in a 1:1 ratio to receive letrozole 2.5 mg or combination of letrozole 2.5 mg and clomiphene 50 mg for 5 days on days 3-7 of menstrual cycle. The women and their partners will be instructed to have regular intercourse with the intent to conceive during the cycle. Patients will have an transvaginal ultrasound mid cycle and to evaluate number of follicles (>15 mm), follicle size, endometrial thickness and pattern. Patients will have mid- luteal phase progesterone level drawn to evaluate ovulation. Side effect profile will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to comply with all study procedures and be available for the duration of the study
2. Diagnosis of infertility: Inability of couple to achieve successful pregnancy after 12 months of regular timed unprotected intercourse in women less than 35 years of age; and after 6 months of regular intercourse without use of contraception in women 35 years and older
3. Diagnosis of polycystic ovary syndrome based on Revised Rotterdam criteria
4. Ability to have regular intercourse during the ovulation induction phase of the study
5. Normal sperm concentration of 15 million/mL and with normal motility of > 40% according to World Health Organization cutoff points, in at least one ejaculate during the previous year

Exclusion Criteria:

1. Current pregnancy
2. Current use of hormonal contraception; use of any type of combined contraceptive or oral progestins within the past month; or use of hormonal implants or depo progestins within the past 3 months
3. Other known cause of infertility: endometriosis, tubal factor, uterine abnormalities
4. Uncorrected thyroid disease
5. Untreated hyperprolactinemia.
6. Medical conditions in which avoiding pregnancy is recommended until under improved control: poorly controlled Type 1 or Type 2 diabetes, poorly controlled hypertension
7. Contraindications to clomiphene citrate: hypersensitivity to CC or any of its components, history of liver disease or known liver disease, unknown cause of abnormal uterine bleeding, or intracranial lesion
8. Contraindications to letrozole: hypersensitivity to letrozole or any of its components.
9. Use of medications known to affect reproductive function or metabolism or that are an absolute contraindication during pregnancy within the past month.
10. If patients are suspected based on clinical findings for other etiologies that mimic PCOS, work up must be completed to exclude other etiologies prior to enrollment (i.e. Cushing's syndrome, androgen-secreting tumor).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Mejia, DO, Principal Investigator — University of Iowa Hosptials & Clinics; Brad Van Voorhis, MD, Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mejia RB, Summers KM, Kresowik JD, Van Voorhis BJ. A randomized controlled trial of combination letrozole and clomiphene citrate or letrozole alone for ovulation induction in women with polycystic ovary syndrome. Fertil Steril. 2019 Mar;111(3):571-578.e1. doi: 10.1016/j.fertnstert.2018.11.030. Epub 2019 Jan 22. PMID 30683591

RESULTS

PARTICIPANT FLOW:
Groups:
- Letrozole: Letrozole 2.5 mg orally for 5 days on cycle days 3-7
  Letrozole
- Letrozole + Clomiphene: Letrozole 2.5 mg orally for 5 days on cycle days 3-7 AND Clomid 50 mg orally for 5 days on cycle days 3-7
  Clomiphene
  Letrozole
Period: Overall Study
Arm/Group | Letrozole | Letrozole + Clomiphene
Started | 35 | 35
Completed | 34 | 33
Not Completed | 1 | 2
Not completed — Pregnancy | 1 | 1
Not completed — Ineliegible due to tuberculosis | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Letrozole + Clomiphene | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (3.9) | 30 (4.4) | 31 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 29 | 30 | 59
  Race/Ethnicity: Black | 2 | 1 | 3
  Race/Ethnicity: Asian | 1 | 1 | 2
  Race/Ethnicity: Hispanic or Latino | 2 | 2 | 4
  Race/Ethnicity: More than 1 race | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33 (8.7) | 34 (7.0) | 33 (7.8)
Weight [Mean (Standard Deviation); unit: kg] | 94 (29.6) | 94 (22.5) | 94 (26.1)
Insurance Coverage [Count of Participants; unit: Participants]
  Full coverage | 10 | 15 | 25
  Partial coverage | 9 | 10 | 19
  No coverage/unsure | 16 | 10 | 26
PCOS Diagnsosis [Count of Participants; unit: Participants]
  Polycystic ovaries according to modified Rotterdam | 35 | 32 | 67
  Hyperandrogenism | 20 | 21 | 41
  Oligomenorrhea | 34 | 33 | 67
Previous Live Birth [Count of Participants; unit: Participants] | 14 | 11 | 25
Duration of Time Attempting to Conceive [Mean (Standard Deviation); unit: months] | 30 (29.6) | 28 (18.5) | 29 (24.5)
Previous use of Letrozole [Count of Participants; unit: Participants] | 10 | 17 | 27
Max dose of Letrzole [Median (Inter-Quartile Range); unit: mg] — Population: Participants who had previously used Letrozole
  mg
    number analyzed (Participants) | 10 | 17 | 27
    (all) | 5 [2.5 to 7.5] | 5 [2.5 to 7.5] | 5 [2.5 to 7.5]
Ovulation on max dose of Letrozole [Count of Participants; unit: Participants] — Population: Participants who had previously used Letrozole.
  Participants
    number analyzed (Participants) | 10 | 16 | 26
    (all) | 4 | 7 | 11
Letrozole use >6 mo before [Count of Participants; unit: Participants] — Population: Participants who had previously used Letrozole.
  Participants
    number analyzed (Participants) | 10 | 16 | 26
    (all) | 6 | 10 | 16
Previous use of Clomiphene [Count of Participants; unit: Participants] | 17 | 23 | 40
Max dose of Clomiphene [Median (Inter-Quartile Range); unit: mg] — Population: Participants who had previously used Clomiphene.
  mg
    number analyzed (Participants) | 17 | 23 | 40
    (all) | 150 [100 to 150] | 150 [100 to 150] | 150 [100 to 150]
Ovulation on max dose of Clomiphene [Count of Participants; unit: Participants] — Population: Participants who had previously used Clomiphene.
  Participants
    number analyzed (Participants) | 16 | 23 | 39
    (all) | 9 | 8 | 17
Clomiphene use >6mo before [Count of Participants; unit: Participants] — Population: Participants who had previously used Clomiphene
  Participants
    number analyzed (Participants) | 16 | 23 | 39
    (all) | 7 | 14 | 21
Previous use of both Letrozole and Clomiphene [Count of Participants; unit: Participants] | 8 | 14 | 22
Resistance to both Letrozole and Clomid [Count of Participants; unit: Participants] — Population: Participants who had previously used both Letrozole and Clomiphene.
  Participants
    number analyzed (Participants) | 8 | 14 | 22
    (all) | 4 | 7 | 11
Metformin Use [Count of Participants; unit: Participants]
  Current Use | 14 | 15 | 29
  Previous Use/Not Current | 6 | 10 | 16
  Never Used | 15 | 10 | 25
HbA1c [Mean (Standard Deviation); unit: mmol/mol] — Population: Participants with prior HbA1c available at baseline.
  mmol/mol
    number analyzed (Participants) | 23 | 23 | 46
    (all) | 5.3 (0.47) | 5.3 (0.73) | 5.3 (0.61)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dL] — Population: Participants who had prior 2-h GTT available.
  mg/dL
    number analyzed (Participants) | 6 | 9 | 15
    (all) | 95 (6.7) | 90 (10.6) | 93 (9.3)
2-hr GTT [Mean (Standard Deviation); unit: mg/dL] — Population: Participants who had prior 2-h GTT available.
  mg/dL
    number analyzed (Participants) | 6 | 9 | 15
    (all) | 103 (18.5) | 114 (23.0) | 110 (21.2)
Current tobacco use [Count of Participants; unit: Participants] | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Ovulation Measured by Mid-luteal Progesterone Level
Description: Ovulation: mid-luteal progesterone > /=3 ng/mL. No ovulation: mid-luteal progesterone <3ng/mL.
Time Frame: 7 days following LH surge or at cycle day 21 if no LH surge was detected
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Letrozole + Clomiphene
Number analyzed (Participants) | 35 | 35
Participants | 15 | 27
Statistical Analysis 1: Comparison: Letrozole vs Letrozole + Clomiphene; Test type: Superiority; p = 0.007, Chi-squared, Corrected; Rate ratio = 1.80, 95% CI 2-sided [1.18 to 2.75]

2. Secondary Outcome: Number of Developing Follicles
Description: Number of follicles measuring > 10mm on ultrasound
Time Frame: Cycle day 12-14
Measure: Median (Inter-Quartile Range); unit: follicles
Arm/Group | Letrozole | Letrozole + Clomiphene
Number analyzed (Participants) | 34 | 33
follicles | 0 [0 to 1] | 1 [0 to 3]
Statistical Analysis 1: Comparison: Letrozole vs Letrozole + Clomiphene; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Size of Largest Developing Follicle
Description: Size of largest follicle on ultrasound
Time Frame: Cycle day 12-14
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Letrozole | Letrozole + Clomiphene
Number analyzed (Participants) | 34 | 33
mm | 10 [8.75 to 15.25] | 16 [10 to 19]
Statistical Analysis 1: Comparison: Letrozole vs Letrozole + Clomiphene; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Endometrial Thickness
Description: Thickness of endometrial lining assessed by ultrasound
Time Frame: Cycle day 12-14
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Letrozole | Letrozole + Clomiphene
Number analyzed (Participants) | 34 | 33
mm | 6.2 (2.2) | 8.3 (3.6)
Statistical Analysis 1: Comparison: Letrozole vs Letrozole + Clomiphene; Test type: Superiority; p = 0.006, t-test, 2 sided

5. Secondary Outcome: Conception
Description: Conception: a positive serum or urinary test of hCG; No conception: Neither a positive serum or urinary test of hCG
Time Frame: 5 weeks after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Letrozole + Clomiphene
Number analyzed (Participants) | 34 | 33
Participants | 3 | 4
Statistical Analysis 1: Comparison: Letrozole vs Letrozole + Clomiphene; This study was not powered to detect significant between-group differences for this conception; Test type: Superiority; p = 0.709, Chi-squared

6. Secondary Outcome: Clinical Pregnancy
Description: Clinical Pregnancy: an intrauterine pregnancy with fetal heart motion determined by ultrasonography; No Clinical Pregnancy: no intrauterine pregnancy with fetal heart motion determined by ultrasonography
Time Frame: 6-7 weeks after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Letrozole + Clomiphene
Number analyzed (Participants) | 34 | 33
Participants | 1 | 3
Statistical Analysis 1: Comparison: Letrozole vs Letrozole + Clomiphene; This study was not powered to detect significant between-group differences for clinical pregnancy; Test type: Superiority; p = 0.356, Chi-squared

7. Secondary Outcome: Multiple Gestation
Description: Multiple Gestation: an intrauterine pregnancy with multiple fetal heart rates determined by ultrasonography; No Multiple Gestation: either no intrauterine pregnancy, or an intrauterine pregnancy with a single fetal heart rate determined by ultrasonography
Time Frame: 9-10 months after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Letrozole + Clomiphene
Number analyzed (Participants) | 34 | 33
Participants | 0 | 0

8. Secondary Outcome: Live Birth
Description: Live Birth: delivery of a live infant; No Live Birth: no delivery of a live infant
Time Frame: 9-10 months after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Letrozole + Clomiphene
Number analyzed (Participants) | 34 | 33
Participants | 1 | 3
Statistical Analysis 1: Comparison: Letrozole vs Letrozole + Clomiphene; This study was not powered to detect significant between-group differences for live birth; Test type: Superiority; p = 0.356, Chi-squared

9. Secondary Outcome: Pregnancy Loss
Description: Pregnancy Loss: any pregnancy loss including biochemical pregnancy, ectopic pregnancy, and miscarriage; No Pregnancy Loss: no pregnancy loss including biochemical pregnancy, ectopic pregnancy, or miscarriage.
Time Frame: 9-10 months after treatment
Population: Participants who conceived
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Letrozole + Clomiphene
Number analyzed (Participants) | 3 | 4
Participants | 2 | 1
Statistical Analysis 1: Comparison: Letrozole vs Letrozole + Clomiphene; This study was not powered to detect significant between-group differences for pregnancy loss; Test type: Superiority; p = 0.486, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Participants were followed for approximately 1 month (1 menstrual cycle) for adverse events related to treatment medication. Participants who became pregnant during the treatment cycle were followed for up to approximately 9 months through the resolution of their pregnancy for adverse events during the pregnancy resulting from the study medication.
Description: Participants were provided with a calendar log to keep track of medication side-effects each day of their treatment cycle. Adverse events in pregnancy were tracked through chart abstraction and participant self reporting.
Arm/Group | Letrozole | Letrozole + Clomiphene
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/32
Other Adverse Events (participants affected / at risk) | 21/33 | 19/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=33) | Letrozole + Clomiphene (N=32)
Gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0) — Gallstones requiring cholecystectomy and hospitalization.
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) — Appendicitis requiring appendectomy and hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=33) | Letrozole + Clomiphene (N=32)
Headache (Nervous system disorders) | 13 | 9
Hot flashes (Reproductive system and breast disorders) | 4 | 10
Abdominal bloating (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Mood changes (Psychiatric disorders) | 1 | 4
Fatigue (General disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1
Breast Discomfort (Reproductive system and breast disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2
Sleep disturbances including insomnia (Psychiatric disorders) | 1 | 2
Abdominal pain including cramps (General disorders) | 6 | 6
Urinary tract infection (Infections and infestations) | 1 | 1
Pilonidal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Echogenic bowel and small head on ultrasound (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Infant born healthy with no birth defects

LIMITATIONS AND CAVEATS:
This study was powered to detect a difference in ovulation rate between the treatment arms. The study was underpowered to detect significant between-group differences for conception, pregnancy, pregnancy loss, and live birth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT02802865/Prot_SAP_000.pdf